CLINICAL TRIAL: NCT02385643
Title: The Efficacy of A Smartphone-based Support System to Reinforce Alcohol Abstinence in Treatment-seeking Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ming-Chyi Huang (Other Government)
Responsible Party: Sponsor-Investigator, Ming-Chyi Huang, Taipei City Hospital, Taipei City Hospital
Organization: Taipei City Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOST 103-2628-B-532 -001 -MY3
Record Dates: First submitted 2015-02-26; First posted 2015-03-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Alcohol Dependence
Keywords: alcohol dependence; abstinence; relapse prevention; mobile support system
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): This group of subjects receives mobile support system and conventional treatment
  Interventions: Behavioral: SmartPhone Support System
- Control group (No Intervention): This group of patients receive conventional treatment only

INTERVENTIONS:
Behavioral: SmartPhone Support System
  Arms: Intervention group

SUMMARY:
Background: Interactive and mobile technology to manage alcohol use problem potentially provide continuing care by offering emotional and instrumental support anywhere and in time, but the effectiveness for maintaining abstinence has not been examined. the investigators will evaluate in this study whether the smartphone-based support system would improve outcomes for people in recovery for alcohol dependence. To enable continuous self-monitoring and self-management, the phone support system prompts subjects to take Breath Alcohol Concentration (BrAC) tests using a phone application and a Bluetooth sensor unit. The system also offers instantaneous feedback, self-management strategies, and anonymous mutual social support from other subjects.

Methods: This three-year project will be conducted in three stages, including pilot study, efficacy evaluation (12 week), and post-intervention follow-up (12 week) stage. Participants will be given a smartphone (if the subject does not have one), breathalyzer and training session. In the pilot study stage,10 subjects will be enrolled to validate the system. In the efficacy evaluation stage, the investigators will conduct a 12-week by enrolling 100 post-detoxification alcohol dependent patients who are randomized to (1) standard treatment (ST) group or (2) standard treatment plus phone-based support group (technology intervention, TI group). Participants will be assessed by Time-Line Follow-Back (TLFB) to record the frequency and quantity of alcohol consumption, visual analogue for craving, Beck Depression Inventory (BDI) and Beck Anxiety Inventory (BAI), Satisfaction with Life Scale (SWLS), and Quality of life Scale (WHOQOL-BREF) and compared for outcome measures. After the 12-week trial, the investigators will take back the support system and follow the all subjects in both groups for another 12 weeks, i.e. post-intervention stage, to further understand the sustaining benefit from intervention. In addition, the investigators will identify the clinical variables or system factors that are associated with outcome measures.

Expected results: In this study, the investigators expect that in treatment-seeking alcohol dependent patients, a smartphone-supported self-management program, adding on to conventional treatment, will be beneficial in improving the drinking outcomes such as a higher abstinence rate, a lower relapse rate, and a lower drinking frequency and quantity.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20 and 50 years;
2. Use an Android phone as his/her primary phone, or be willing to use an Android phone provided by National Taiwan University as his/her primary phone during the study;
3. Fulfilling the Diagnostic and Statistical Manual version IV (DSM-IV) criteria of alcohol dependence assessed by the Structured Clinical Interview;
4. Complete abstinence for at least 10 days and free of any withdrawal symptoms; and
5. Drug screening test results negative opiates, amphetamines, and ketamine.

Exclusion Criteria:

1. A current DSM-IV diagnosis of dependence or abuse on other substances except nicotine or the use of one to two low-potency benzodiazepine tablets for sleep impairment;
2. A current mental or psychiatric impairment or disease that required psychotropic medication or inpatient treatment on a psychiatric ward;
3. A history of opioid or psychostimulant abuse;
4. A history of psychosis, including schizophrenia, bipolar I or bipolar II disorder, and major depressive disorder with psychotic features;
5. Current use of any antipsychotics;
6. Homelessness;
7. Pregnancy, nursing, or refusal to use a reliable method of birth control in women;
8. Cognitive deficit and not thus being able to comprehend the informed consent and study procedure

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-09; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Time to first lapse | 12 weeks
Time to first relapse | 12 weeks
Cumulative abstinence days | 12 weeks
Number of drinks per drinking days | 12 weeks
  each visit during the 12 weeks: week 1, 2, 4, 8, 12
VAS craving measurement | 12 weeks
  each visit during the 12 weeks: week 1, 2, 4, 8, 12
complete abstinence rate | 12 weeks
Drop-out rate | 12 weeks
  each visit during the 12 weeks: week 1, 2, 4, 8, 12

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Chyi Huang, MD, PhD, Principal Investigator — Taipei City Psychiatric Center; Hao-Hua Chu, PhD, Study Chair — Department of Computer Science and Information Engineering, National Taiwan University; Chuang-Wen You, PhD, Study Director — Intel-NTU Connected Context Computing Center, National Taiwan University
Locations (1):
- Ming-Chyi, Taipei, Taiwan